CLINICAL TRIAL: NCT00209105
Title: Emory Conte Center for the Neuroscience of Mental Disorders: Psychobiology of Childhood Trauma
Brief Title: Characterizing Psychological Consequences of Childhood Trauma
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Becky Kinkead, PhD, Assocate Professor, Emory University
Other Study IDs: IRB00021800; P50MH058922 (NIH); 572-2004; DATR A3-NSC
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Major Depressive Disorder
Keywords: Child Abuse; Hypothalamic-Pituitary-Adrenal Axis; Brain Imaging; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Participants who have experienced early-life trauma will undergo a series of diagnostic tests.
  Interventions: Drug: DEX-CRF stimulation test; Behavioral: Psychosocial stress induction; Procedure: Brain imaging of sad mood , self-reference, reward; Behavioral: Acoustic startle

INTERVENTIONS:
Drug: DEX-CRF stimulation test — 1 ug/kg body weight of CRF for determining hpa response post dexamethasone ingestion
Behavioral: Psychosocial stress induction — Laboratory stress induction, no drug administration
Procedure: Brain imaging of sad mood , self-reference, reward — Brain imaging
Behavioral: Acoustic startle — No drugs involved

SUMMARY:
This study will characterize the mental health consequences of early-life trauma.

DETAILED DESCRIPTION:
This primary goal of this Center is to characterize the neurobiological consequences of early-life trauma. The Center comprises 6 projects that include human subjects. Human subjects are recruited through Project 6.

Project 2: Psychoimmunology (PI A.H. Miller) Project 4: A Model of Learned Safety(PI: M. Davis) Project 6: Clinical Psychobiology(PI: C. Heim) Project 7: Children of Depressed Mothers(PI: Z. Stowe) Project 8: Functional Brain Imaging (PIs: H.S. Mayberg, G. Berns) Project 9: Structural & Anatomical Connectivity Studies (PI: C.Kilts, X. Hu).

Project 2: The study seeks to examine the impact of psychosocial stress on neuroendocrine and immune signaling pathways of adult men and women with and without major depression who have experienced serious trauma (abuse, loss) during development. Serial blood samples will be collected at baseline and after an acute speech/math stressor (see Project 6). Assessments include IL-1alpha, and beta, IL-6, TNF alpha as well as DNS binding of relevant neuroendocrine-immune transcription factors, i.e. GR, CREB, and NFkB.

Project 4: This study uses a model of that allows for the independent evaluation of excitation and inhibition of fear-conditioning measured with the acoustic startle reflex. In addition, a dark-enhanced startle paradigm will be used that tests for anxiety. The effects of early-life stress will be evaluated in humans with and without major depressive disorder.

Project 6: This study assesses neuroendocrine and autonomic responses to stress and pharmacological challenge in subjects with and without major depression who have or have nor experienced early life stress. We seek to identify causes of variability in neuroendocrine-autonomic outcome after early life stress. To achieve this principle aim, we study the role of moderating and mediating factors including gender, genotype, type/timing of childhood trauma, as well as the role of adulthood trauma, comorbidity and cognitive dysfunction. The projects serves as a human subjects core for the other projects.

Project 7: This project characterizes effects of maternal depression on offspring in a longitudinal study. Women with and without depression will be prospectively followed through pregnancy and the first 6 months post-partum. Maternal stress and psychopathology, pregnancy and birth complications, medications and infants' physiological and behavioral stress responses will be assessed.

Project 8: This study uses PET and fMRI to characterize the impact of early-life stress on functional neural pathways mediating mood reactivity, self reference and reward-processing in patients with major depression. Cortical-limbic-striatal changes in cases with early stress but no psychopathology that define vulnerability to depression are also identified.

Project 9: This Project uses data obtained in Project 8 as well as diffusion tensor imaging to define the influence of early-life trauma on brain anatomical and functional connectivity.

ELIGIBILITY:
Inclusion Criteria:

* For participants assigned to the MDD groups: current DSM-IV diagnosis of MDD
* For participants assigned to the early-life stress group: repeated (once per month or more for at least year) sexual or physical abuse before the age of 13 years by a perpetrator at least 5 years older at the time
* For female participants: regular menstrual cycle and assessment in the early follicular phase as verified by sex steroid measures

Exclusion Criteria:

* Meets DSM-IV criteria for a gender identity disorder
* For all participants assigned to non-MDD groups: DSM-IV diagnosis of current MDD
* For all participants assigned to the group without early-life stress: major stress experiences before the age of 12 years, such as separation from parents, neglect, parental loss, accidents, severe illness, or natural disaster
* Significant medical illness, such as gastrointestinal, neurological, hormonal, heart, lung, kidney, liver, immunological or hematological disease, organic brain disease, or cancer as determined by history, physical examination, ECG, and laboratory tests
* Pregnant or breastfeeding
* Past or current presence of psychotic symptoms or bipolar disorder
* Current presence of psychoactive substance abuse/dependency or eating disorders
* Currently taking hormonal medication
* Taking psychotropic medication within 4 weeks of study entry
* General exclusion criteria for PET and fMRI

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will include participants who have experienced early-life trauma.
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2005-01; Primary Completion 2009-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Pathophysiological pathways (e.g., blood chemicals, physiological measures, brain images, behavioral measures), as assessed by diagnostic tests | Measured at Day 2.5

CONTACTS AND LOCATIONS:
Overall Officials: Becky Kinkead, PhD, Principal Investigator — Emory University SOM - Dept. of Psychiatry and Behavioral Sciences
Locations (1):
- General Clinical Research Center at Emory University Hospital, Atlanta, Georgia, United States